CLINICAL TRIAL: NCT02275351
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Vehicle- Controlled Study of the Safety, Tolerability, and Efficacy of 0.15% and 0.25% Concentrations of Topical SM04554 Solution in Male Subjects With Androgenetic Alopecia (AGA)
Brief Title: A Study of the Safety, Tolerability, and Efficacy of Topical SM04554 Solution in Male Subjects With Androgenetic Alopecia (AGA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SM04554-AGA-02
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Androgenetic Alopecia
Keywords: alopecia; topical; Samumed
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active Arm 1 (Experimental): Topical SM04554 0.15% solution, applied once a day for 90 days
  Interventions: Drug: SM04554
- Active Arm 2 (Experimental): Topical SM04554 0.25% solution, applied once a day for 90 days
  Interventions: Drug: SM04554
- Vehicle Arm (Placebo Comparator): Topical vehicle solution, applied once a day for 90 days
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: SM04554 — Topical solution, applied once a day
  Arms: Active Arm 1; Active Arm 2
Drug: Vehicle — Topical solution, applied once a day
  Arms: Vehicle Arm

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, and efficacy of topical SM04554 solution (0.15% and 0.25%) applied to the scalp of male subjects with Androgenetic Alopecia (AGA).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of AGA
* Willing to inform females, with whom they may interact, that they are using a topical investigational product and direct contact should be avoided as potential harm to a fetus is unknown
* Willing to maintain the same hair style as at study start for the duration of the study
* Willing to not use semi-permanent hair products (e.g., color, texturizers, relaxers) for the duration of the study. Daily styling products will be allowed (e.g., hair gel, mousse, styling spray).
* Willing to use a mild non-medicated shampoo and conditioner for the duration of the study
* Willing to receive a small scalp tattoo
* Able to read and understand English

Exclusion Criteria:

* Clinical diagnosis of alopecia areata or other non-AGA forms of alopecia
* Scalp hair loss on the treatment area, due to disease, injury, or medical therapy
* Males who are sexually active and have a partner who is capable of becoming pregnant, neither of whom have had surgery to become sterilized, that are not using an effective method of birth control and are not willing to use an effective method of birth control during the study treatment period until 90 days post last dose of study medication
* Current skin disease (e.g., psoriasis, atopic dermatitis, skin cancer, eczema, sun damage, seborrheic dermatitis), cuts and/or abrasions on the scalp or condition (e.g., sunburn, tattoos) on the treatment area that, in the opinion of the Investigator, might put the subject at risk or interfere with the study conduct or evaluations
* History of surgical correction of hair loss on the scalp
* Previous exposure to SM04554
* Use of any products or devices purported to promote scalp hair growth (e.g., finasteride or minoxidil) within the 24 weeks prior to study start
* Use of anti-androgenic therapies (e.g., spironolactone, flutamide, cyproterone acetate, cimetidine) within 12 weeks prior to study start
* History of hair transplants
* Current use of an occlusive wig, hair extensions, or hair weaves
* Participation in any other investigational drug or medical device trial, which included administration of an investigational study medication or medical device, within 30 days or 5 half-lives of the investigational agent, whichever is longer, prior to study start
* Subjects with a history of clinically significant cardiac arrhythmia as determined by the Investigator
* Subjects with clinically significant findings from medical history, clinical laboratory tests, electrocardiogram (ECG), or vital signs that, in the opinion of the Investigator, could interfere with the objectives of the study or put the subject at risk
* Subjects unwilling to refrain from sperm donation during the study treatment period until 90 days post last dose of study medication
* Subjects with pregnant partners at study start
* Use of semi-permanent hair products (e.g., color, texturizers, relaxers) within 30 days prior to study start
* Use of medicated shampoo or conditioner within 30 days prior to study start

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 310 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in non-vellus hair count | Baseline, Day 45, Day 90
  Change in non-vellus hair count over time as compared to Baseline. Non-vellus hair count will be determined by macrophotography.
Change in subject assessment of hair growth and quality | Day 45, Day 90
  Change in Men's Hair Growth Questionnaire (MHGQ) over time as compared to Baseline. The MHGQ is a subject-completed assessment that asks the subject to evaluate his hair growth and quality since the start of the study.

SECONDARY OUTCOMES:
Change in hair growth as assessed by the investigator | Day 45, Day 90
  Change in hair growth over time as compared to Baseline, as assessed by the investigator, using a 7-point scale from -3 (greatly decreased) to +3 (greatly increased).
Impact of AGA on quality of life | Baseline, Day 45, Day 90
  Change in subject responses to the Kingsley Alopecia Profile (KAP) questionnaire over time as compared to Baseline. The KAP is a 38-question survey completed by each subject that assesses his quality of life in relation to AGA.
Change in hair density | Baseline, Day 45, Day 90
  Change in hair density over time as compared to Baseline. Hair density will be measured using macrophotography.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, M.D., Study Director — Biosplice Therapeutics, Inc.
Locations (23):
- United States (23):
  - Encinitas, California
  - San Diego, California
  - New Haven, Connecticut
  - Miami, Florida
  - West Palm Beach, Florida
  - Plainfield, Indiana
  - Wichita, Kansas
  - Clinton Township, Michigan
  - Detroit, Michigan
  - Fridley, Minnesota
  - Albuquerque, New Mexico
  - New York, New York
  - Stony Brook, New York
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Portland, Oregon
  - Austin, Texas
  - College Station, Texas
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Lynchburg, Virginia
  - Norfolk, Virginia